CLINICAL TRIAL: NCT00769600
Title: A Randomized Phase II Study of Itraconazole and Pemetrexed in Patients With Previously Treated Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Phase II Study of Itraconazole and Pemetrexed in Patients With Previously Treated Non-Squamous NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0881JS; NA_00020074 (Other: Johns Hopkins Institutional Review Board 2)
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Recurrent Non Small Cell Lung Cancer
Keywords: Recurrent Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Itraconazole; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Itraconazole with Pemetrexed (Active Comparator): Pemetrexed IV every 21 days with oral Itraconazole 200mg daily.
  Interventions: Drug: Itraconazole; Drug: Pemetrexed
- Single agent pemetrexed (Active Comparator): Pemetrexed IV on day 1 of 21-day cycle.
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Itraconazole — Itraconazole 200 mg once daily
  Other Names: Sporanox
  Arms: Itraconazole with Pemetrexed
Drug: Pemetrexed — Pemetrexed every 21 days.
  Other Names: Alimta

SUMMARY:
Primary Objective

To evaluate the 3-month event-free survival of the combination of the combination of itraconazole and pemetrexed in patients with recurrent/refractory non-small cell lung cancer.

Secondary Objectives

To determine the objective response rate of the combination of itraconazole and pemetrexed in patients with recurrent/refractory non-small cell lung cancer.

DETAILED DESCRIPTION:
Primary Objective

To evaluate the 3-month event-free survival of the combination of the combination of itraconazole and pemetrexed in patients with recurrent/refractory non-small cell lung cancer. 3-month event-free survival (EFS) is defined as the proportion of patients who are alive and without event after 3 months (evaluated in a window of +/- 1 week) of treatment. Events are defined as disease progression or death from any cause. All patients treated on protocol will be included in the determination of EFS, regardless of treatment modification or discontinuation.

Secondary Objectives

To determine the objective response rate of the combination of itraconazole and pemetrexed in patients with recurrent/refractory non-small cell lung cancer. The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for progressive disease the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed NSCLC.
* Patient must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 11 for the evaluation of measurable and non-measurable disease.
* Patients must have received at least one previous chemotherapy regimen and have recurrent or refractory disease.
* Age >18 years. Because no dosing or adverse event data are currently available on the use of itraconazole in combination with pemetrexed in patients < 18 years of age, such patients are excluded from this study but will be eligible for future pediatric phase 2 combination trials.
* Life expectancy of greater than 12 weeks.
* ECOG performance status < 2 (Karnofsky > 60%; see Appendix A).
* Patients must have normal organ and marrow function as defined below:

  * leukocyte > 3,000/mcL
  * absolute neutrophil count > 1,500/mcL
  * platelets > 100,000/mcL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT)< 2.5 X institutional upper limit of normal
  * creatinine within normal institutional limits
  * creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier.
* Patients may not be receiving any other investigational agents.
* Patients who have received prior pemetrexed chemotherapy.
* Patients with uncontrolled brain metastases. Patients with brain metastases must have stable neurologic status following local therapy (surgery or radiation) for at least 2 weeks, and must be without neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to itraconazole and pemetrexed or other agents used in the study.
* Itraconazole is a strong CYP3A4 inhibitor and may increase plasma concentrations of drugs metabolized by this pathway. Coadministration of cisapride, midazolam, pimozide, quinidine, lovastatin, simvastatin, triazolam, dofetilide, or levacetylmethadol (levomethadyl) with itraconazole is contraindicated. Patients who take any of these medications and who are not able to change to an alternative medication will be excluded. Lists including medications and substances known or with the potential to interact with the CYP3A4 isoenzymes are provided in Section 7.1.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because itraconazole and pemetrexed are Class C and D agents, respectively, with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with itraconazole and pemetrexed, breastfeeding should be discontinued if the mother is treated with itraconazole or pemetrexed. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with itraconazole or pemetrexed. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2008-11; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles M Rudin, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States
- Singapore General Hospital, Tiong Bahru Estate, Singapore

REFERENCES:
- [Result] Rudin CM, Brahmer JR, Juergens RA, Hann CL, Ettinger DS, Sebree R, Smith R, Aftab BT, Huang P, Liu JO. Phase 2 study of pemetrexed and itraconazole as second-line therapy for metastatic nonsquamous non-small-cell lung cancer. J Thorac Oncol. 2013 May;8(5):619-23. doi: 10.1097/JTO.0b013e31828c3950. PMID 23546045

RESULTS

PARTICIPANT FLOW:
Groups:
- Itraconazole Open Label Added to Standard of Care Pemetrexed: Subjects will receive standard dose pemetrexed day 1 of each 21-day cycle, IV. Participants will be randomized at the beginning of the study to receive either oral itraconazole 200 mg once daily during the period of chemotherapy (days 1-21).
  Itraconazole: Itraconazole 200 mg once daily
- Single Agent Pemetrexed: Subjects will receive standard dose pemetrexed day 1 of each 21-day cycle, IV. Participants will be randomized at the beginning of the study to receive pemetrexed alone.
  Pemetrexed
Period: Overall Study
Arm/Group | Itraconazole Open Label Added to Standard of Care Pemetrexed | Single Agent Pemetrexed
Started | 15 | 8
Completed | 15 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Itraconazole Open Label Added to Standard of Care Pemetrexed | Single Agent Pemetrexed | Total
Number analyzed (Participants) | 15 | 8 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 5 | 17
  >=65 years | 3 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 60 [49 to 75] | 59 [48 to 72] | 59.5 [48 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 8 | 3 | 11
Region of Enrollment [Number; unit: participants]
  United States | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Median number of days alive
Time Frame: up to 3 years
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Arm A: Itraconazole plus pemetrexed
- Arm B: Pemetrexed alone
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 15 | 8
days | 971 [426 to 1135] | 242 [128 to NA] — the upper limit is not reached due to small sample size

2. Primary Outcome: Progression Free Survival as Measured by Number of Days Without Disease Progression
Time Frame: 1 year
Measure: Median (Full Range); unit: days
Groups:
- Single Agent Pemetrexed: Subjects will receive standard dose pemetrexed day 1 of each 21-day cycle, IV. Participants will be randomized at the beginning of the study to receive pemetrexed alone.
Arm/Group | Itraconazole Open Label Added to Standard of Care Pemetrexed | Single Agent Pemetrexed
Number analyzed (Participants) | 15 | 8
days | 168 [82 to 364] | 84 [21 to 210]

3. Primary Outcome: RECIST Response
Description: Number of participants with partial response (PR), stable disease (SD) and progressive disease (PD) as defined by Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: Up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Itraconazole Open Label Added to Standard of Care Pemetrexed | Single Agent Pemetrexed
Number analyzed (Participants) | 15 | 8
Participants
  PR | 3 | 0
  SD | 8 | 5
  PD | 2 | 2
  Inevaluable | 2 | 1

4. Secondary Outcome: Tumor Blood Flow
Description: Tumor blood flow activity in patients with previously treated non-squamous non-small cell lung cancer receiving pemetrexed alone or pemetrexed plus itraconazole.
Time Frame: 3 years
Population: Data was not collected to assess this outcome measure.
Arm/Group | Itraconazole Open Label Added to Standard of Care Pemetrexed | Single Agent Pemetrexed
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Tumor Metabolic Activity
Description: Tumor metabolic activity in patients with previously treated non-squamous non-small cell lung cancer receiving pemetrexed alone or pemetrexed plus itraconazole.
Time Frame: 3 years
Population: Data was not collected to assess this outcome measure.
Arm/Group | Itraconazole Open Label Added to Standard of Care Pemetrexed | Single Agent Pemetrexed
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: up to 30 days post last treatment.
Arm/Group | Itraconazole Open Label Added to Standard of Care Pemetrexed | Single Agent Pemetrexed
All-Cause Mortality (participants affected / at risk) | 6/15 | 6/8
Serious Adverse Events (participants affected / at risk) | 2/15 | 2/8
Other Adverse Events (participants affected / at risk) | 3/15 | 2/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole Open Label Added to Standard of Care Pemetrexed (N=15) | Single Agent Pemetrexed (N=8)
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Pulmonary Embolus (Cardiac disorders) | 0 | 1
Intratumoral Bleed (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Itraconazole Open Label Added to Standard of Care Pemetrexed (N=15) | Single Agent Pemetrexed (N=8)
Lymphopenia (Blood and lymphatic system disorders) | 3 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vertigo (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No